CLINICAL TRIAL: NCT02862834
Title: Towards an Improvement in Diagnosis and Genetic Counselling in Syndromic Poikiloderma
Brief Title: Screening for Genes in Patients With Poikiloderma
Acronym: poikiloderma
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Courcet AOI 2012
Record Dates: First submitted 2016-08-05; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Poikiloderma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with poikiloderma
  Interventions: Genetic: High-throughput exome sequencing

INTERVENTIONS:
Genetic: High-throughput exome sequencing

SUMMARY:
In the context of this study, the investigators wish to take advantage of high-throughput genetic techniques (microarray and high-throughput exome sequencing) to identify new genes implicated in syndromic poikiloderma so as to improve the diagnostic decision tree in these syndromes, opportunities for genetic counselling for patients and their families and the follow-up of patients, notably with regard to the risk of tumours.

This study will make it possible to identify new genes implicated in syndromic poikiloderma and improve the diagnostic strategy proposed to patients with these syndromes, and to propose to patients a confirmed diagnosis, appropriate follow-up, notably with regard to the risk of tumours, genetic counselling to families and eventually an antenatal diagnosis to couples who would like to have one for future pregnancies.

The identification of new genetic causes of syndromic poikiloderma will also make it possible to complete the current classification of these syndromes

ELIGIBILITY:
Inclusion Criteria:

patients with syndromic poikiloderma, defined by the association of poikiloderma with other extradermatological clinical signs,

* normal array-CGH, screening for chromosomal rearrangements,
* absence of mutations in the genes RECQL4, KIND1 or C16orf57,
* sporadic or familial involvement.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with poikiloderma
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Identification of novel genes involved in syndromic poikiloderma | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France